CLINICAL TRIAL: NCT05972460
Title: IMM2510, a Multi-Center, Open-Label, Dose Escalation and Cohort Expansion Phase I Clinical Study for Advanced Solid Tumors
Brief Title: IMM2510, a PD-L1 and VEGF Bispecific Fusion Protein, in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM2510-01
Record Dates: First submitted 2023-03-27; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM2510 in Advanced Solid Tumors (Experimental): IMM2510 Phase 1a Dose Escalation: 0.007 mg/kg, 0.03 mg/kg, 0.1 mg/kg, 1.0 mg/kg, 3.0 mg/kg, 6.0 mg/kg, 10 mg/kg, 20 mg/kg, or higher dose, through intravenous administration every 2 weeks up to 52 weeks.
  Phase 1b Cohort Expansion: multiple cohorts are planned, including, but not limited to: non-small cell lung cancer, liver cancer, cervical cancer, cholangiocarcinoma, pancreatic cancer and renal cell carcinoma, with at least 12 patients enrolled in each cohort to further explore the safety and efficacy of IMM2510 in different tumors. The dose for expansion is given by intravenous infusion up to 52 weeks.
  Interventions: Drug: IMM2510

INTERVENTIONS:
Drug: IMM2510 — IMM2510 is administered intravenously every 2 weeks, every 28 days for a treatment cycle.
  Other Names: IMM2510 Injection

SUMMARY:
This trial is a first-in-human, open-label, multi-center, dose escalation phase 1a study followed by cohort expansion phase 1b study to evaluate the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of IMM2510, a PD-L1 and VEGF bispecific fusion protein, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
IMM2510 is administered via intravenous infusion every 2 weeks up to 52 weeks. Phase 1a Dose Escalation: using accelerated titration followed by 3+3 dose escalation design to explore the maximum tolerated dose (MTD) and the recommended dose (RDE). Phase 1b Cohort Expansion: planing to enroll at least 60 patients with different advanced solid tumors (multiple cohorts) to further observe the safety and antitumor activity of IMM2510, and to determine the recommended phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily sign the informed consent form; they were able to communicate well with the investigator and comply with the study requirements.
2. Age ≥ 18 years old.
3. Advanced solid tumors confirmed by histology or cytology, failed standard therapy, no standard therapy, or unable to tolerate current standard therapy.
4. Presence of at least one measurable tumor lesion (according to RECIST 1.1 criteria), defined as the maximum longest diameter of 10 mm for imaging (CT/MRI) or 15 mm for a single pathological lymph node lesion; the presence of at least one evaluable tumor lesion is allowed in the dose escalation phase.
5. Life expectancy of at least 3 months.
6. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
7. Organ or bone marrow function must meet the following criteria:

   1. Hematology (no blood component or cell growth factor was used to support therapy within 7 days prior to study treatment): absolute neutrophil count ≥ 1.5×109/L; Hemoglobin ≥ 90 g/L; Platelet count ≥ 100×109/L.
   2. Serum total bilirubin ≤ 1.5× upper limit of normal (ULN) (unless Gilbert syndrome is confirmed); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; ALT and AST were ≤ 5.0×ULN when the elevation was judged to be due to liver metastasis.
   3. Prothrombin time (PT) ≤ 1.2×ULN, partial prothrombin kinase time (APTT) ≤ 1.2×ULN; International Standardized ratio (INR) ≤ 1.2 (unless receiving warfarin treatment); After 2 weeks of oral anticoagulant therapy, the dose is stable. If warfarin is taken orally, the patient must have an INR ≤ 2.5 and no bleeding.
   4. Endogenous creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula), urinary protein < 2+ or protein quantity < 1.0 g.
   5. Left ventricular ejection fraction (LVEF) ≥50%.
8. Toxicity of previous treatment has been restored to grade 1 [NCI CTCAE 5.0 grading standard was adopted] (except for hair loss and chemotherapy-induced neurotoxicity ≤ grade 2 and other toxicity judged by researchers to be without safety risk).
9. Women and men of childbearing age must agree, after signing an informed consent form, to use effective contraception during the study period and within three months after the final dose, and women of childbearing age must have a negative pregnancy test result 72 hours before the dose.
10. The patient is willing and able to comply with protocol visits, treatment protocols, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. Enrol in another clinical study at the same time, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study.
2. Received the last systemic antitumor therapy, including chemotherapy, immunotherapy, and biological agents, within 3 weeks before the first administration; Received hormone antitumor therapy and small-molecule targeted therapy within 2 weeks before the first administration; Palliative local therapy was performed for non-target lesions within 2 weeks before the first administration; Nonspecific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor, not IL-11 for thrombocytopenia) was administered within 2 weeks prior to initial administration; Received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week prior to initial administration.
3. Patients with active central nervous system (CNS) metastasis, but the following patients were admitted: a. Treated patients with brain metastases (such as surgery and radiotherapy), stable for at least 2 weeks after treatment (before the first administration of the study drug), no evidence of new metastatic lesions or metastatic lesion enlargement, and corticosteroid withdrawal ≥3 days before the study drug administration; b. Untreated, asymptomatic subjects with brain metastases who do not require corticosteroids and whose brain metastases are no more than 1.5 cm in length.
4. Receiving >1 programmed cell death protein-1 (PD-1) and its ligand (PD-L1) inhibitors, such as pembrolimab, opdivo, Atzumab, or Devarumab, or > 1 anti-angiogenesis inhibitor, such as bevacizumab, ramolumab, Apatinib, or Regofenib; Or received PD-1/PD-L1 inhibitors and antiangiogenic inhibitors at the same time (including different time sequences of therapy).
5. Developed other malignant tumors within 5 years prior to enrollment. Exceptions: 1) cured cervical carcinoma in situ and non-melanoma skin cancer; 2) Patients with radical treatment, unless they had a complete response for at least 2 years prior to enrollment and did not require additional treatment or did not require additional treatment during the study period.
6. Active, known secondary primary cancer that has not recurred within five years; Exceptions: 1) Both primary and secondary cancers were considered to benefit from this study; 2) The investigators have clearly ruled out which primary tumor source the metastases belong to.
7. History of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disease, multiple sclerosis, etc. Except the following diseases, they are allowed to be included in the group:

   * Hypothyroidism that can be controlled with hormone replacement therapy alone
   * Skin diseases that do not require systemic treatment (e.g. Vitiligo, psoriasis)
   * Celiac disease under control.
8. Patients who had received major surgery within 4 weeks before enrollment; Had received minor surgical procedures (including catheterization, but not peripheral venipuncture central venous catheterization) within 2 days before enrollment.
9. High blood pressure that medications fail to control (systolic blood pressure 140mmHg and/or diastolic blood pressure 90mmHg) or pulmonary hypertension or unstable angina pectoris; Previous myocardial infarction or bypass grafting or stent surgery within 6 months prior to drug administration; History of chronic heart failure with the New York Heart Association (NYHA) criteria of Grade 3-4; Clinically significant valvular disease; Severe arrhythmias requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia), Including QTcF 450ms for men and 470ms for women (calculated by Fridericia formula); Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 months before enrollment.
10. History of arterial thrombosis, deep vein thrombosis and pulmonary embolism within 6 months prior to enrollment.
11. Patients with skin wounds, surgical sites, wound sites, mucous membrane ulcers or fractures that are not fully healed were judged by the researchers to be at risk of bleeding when participating in the study.
12. Conditions that may cause bleeding or perforation of the digestive tract (e.g. duodenal ulcer, intestinal obstruction, acute Crohn's disease, ulcerative colitis, extensive removal of the stomach and small intestine, etc.); Patients with chronic Crohn's disease and ulcerative colitis (except for total colon and rectal excision) should be excluded even during inactive periods; Hereditary nonpolyposis colorectal cancer or familial adenomatous polyposis syndrome; Patients with past history of intestinal perforation and intestinal fistula, but not cured after surgical treatment; Esophageal and gastric varices.
13. Present or past symptoms of idiopathic pulmonary fibrosis or idiopathic pneumonia; Acute lung disease, interstitial lung disease or pneumonia (except local interstitial pneumonia induced by radiotherapy), pulmonary fibrosis, etc.; Patients with severe dyspnea, pulmonary insufficiency or continuous oxygen inhalation.
14. Uncontrolled fluid with repeated drainage or obvious symptoms in the chest, abdomen and pericardium.
15. Subjects who required systemic corticosteroid (dose equivalent to > 10 mg/day of prednisone) or other immunosuppressive drug treatment within 14 days prior to enrollment or during the study period; The following conditions allow inclusion:

    * Subjects are permitted to use topical or inhaled corticosteroids
    * Short-term (≤ 7 days) use of glucocorticoids is permitted for the prevention or treatment of non-autoimmune allergic diseases
16. Patients who were severely infected within the first 4 weeks of enrollment, or who had any signs or symptoms of active infection within the first 2 weeks, or who required antibiotic therapy within the first 2 weeks (except for prophylactic antibiotics); Unexplained fever > 38.5℃ before the first administration (the subjects could be enrolled if their fever was due to tumor, according to the investigators).
17. People infected with active tuberculosis.
18. History of organ transplantation or hematopoietic stem cell transplantation.
19. History of human immunodeficiency virus (HIV) infection or other acquired or congenital immunodeficiency diseases.
20. Hepatitis B surface antigen (HBs-Ag) positive, and HBV-DNA ≥ 2000 IU/mL or beyond the normal line; Hepatitis C (HCV) ribonucleic acid (RNA) positive.
21. Attenuated vaccine is expected to be given 4 weeks before administration, during treatment or within 30 days of the last administration.
22. Patients with previous severe allergic reactions to macromolecular protein preparations/monoclonal antibodies.
23. Permanent discontinuation of the drug due to immune-related toxicity during previous antitumor immunotherapy.
24. Poor compliance with a clear past history of neurological or psychiatric disorders, such as epilepsy, dementia, or alcohol, drug or substance abuse.
25. Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
AEs | From the first dose to 60 days after the last dose of IMM2510, all patients included
  Incidence and characteristics of adverse events (AEs), including serious adverse events (SAEs).
DLT | During 28 days after the first dose of IMM2510, all patients included
  Incidence and characteristics of dose limiting toxicity (DLT).
MTD and RP2D | All patients complete the safety evaluation and confirm the efficacy assessment, up to 52 weeks of treatment per patient
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of IMM2510 in patients with advanced solid tumors.
Changes in Laboratory Test Result | From the first dose to 60 days after the last dose of IMM2510, all patients included
  Changes of blood routine, clinical biochemistry, urine routine, stool routine, coagulation function, thyroid function and other indexes after patients treated with investigational drug compared with those before treatment.
Changes in Electrocardiogram | From the first dose to 60 days after the last dose of IMM2510, all patients included
  Changes in electrocardiogram indicators (heart rate, RR interval, PR interval, QT interval, QRS wave, QT interval, etc.) of patients relative to baseline.
Changes in Vital Signs | From the first dose to 60 days after the last dose of IMM2510, all patients included
  Changes in vital signs (including temperature, blood pressure, breathing, pulse) of patients relative to baseline.
Changes in Physical Examination | From the first dose to 60 days after the last dose of IMM2510, all patients included
  Changes in physical examination (including general conditions, skin, lymph nodes, eyes, ears, nose, mouth, throat, neck, thyroid, chest, lungs, cardiovascular, abdominal, limbs, musculoskeletal and specialist examinations) of patients relative to baseline.

SECONDARY OUTCOMES:
ORR | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Objective Response Rate (ORR) is the proportion of patients with complete response (CR) or partial response (PR). ORR and other efficacy evaluation indexes were based on RECIST 1.1 criteria.
DOR | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Duration of Response (DOR) is the time between the first onset of CR or PR and the first onset of disease progression (PD) or death from any cause. For patients with unknown progression or death, the time of sustained remission was censored at the time point of the last patient evaluation.
DCR | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Disease control rate (DCR) is the proportion of patients with CR, PR, and stable disease (SD).
PFS | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Progression-free survival (PFS) is the time between first initiation of study treatment to PD or death due to any reason. For patients with unknown progression or death, disease-free survival was censored at the time point of the last patient evaluation.
  Duration of Response (DOR) DOR is the time between the first onset of CR or PR and the first onset of disease progression (PD) or death from any cause. For patients with unknown progression or death, the time of sustained remission was censored at the time point of the last patient evaluation.
  Disease control rate (DCR) DCR is the proportion of patients with complete response (CR), partial response (PR), and stable disease (SD).
  Progression-free survival (PFS) PFS is the time between first initiation of study treatment to disease progression (PD) or death due to any reason. For patients with unknown progression or death, disease-free survival was censored at the time point of the last patient evaluation.
Tmax | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Peak time (Tmax), in single dose period and multiple administration periods.
T1/2 | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Elimination phase half-life (T1/2), in single dose period and multiple administration periods.
Cmax | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Peak concentration (Cmax), in single dose period.
AUC0-tlast | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Area under plasma concentration-time curve from 0 to the last quantifiable time point (AUC0-tlast), in single dose period.
AUC0-inf | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Area under plasma concentration-time curve from 0 to infinite time (AUC0-inf), in single dose period.
V | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Volume of distribution (V), in single dose period.
CL | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Clearance (CL), in single dose period.
Cmin, ss | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Steady-state trough concentration (Cmin, ss), in multiple administration periods.
Cmax, ss | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Steady-state peak concentration (Cmax, ss), in multiple administration periods.
Cav, ss | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Mean plasma concentration at steady state (Cav, ss), in multiple administration periods.
AUC0-tau | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Area under the drug-time curve (AUC0-tau), in multiple administration periods.
Rac _ Cmax | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Cmax accumulation ratio (Rac _ Cmax), in multiple administration periods.
Vss | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  Steady-state distribution volume (Vss), in multiple administration periods.
CLss | From IMM2510 dosing of the first patient to the last patient completing a maximum of 52 weeks of treatment
  steady-state clearance (CLss), in multiple administration periods.

CONTACTS AND LOCATIONS:
Overall Officials: Qiying Lu, MD, Study Director — ImmuneOnco Biopharmaceuticals (Shanghai) Inc.
Locations (4):
- China (4):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Shandong Provincial Institute of Cancer Prevention and Treatment, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No